CLINICAL TRIAL: NCT02862873
Title: Iinterest of Intravenous Ondansetron in the Prevention of Spinal Anaesthesia-induced Hypotension in Caesarean Section: Double-blind Randomized Controlled Single-centre Study
Brief Title: Interest of Intravenous Ondansetron in the Prevention of Spinal Anaesthesia-induced Hypotension in Caesarean Section
Acronym: ZORA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GIRARD WOLFF 2014
Record Dates: First submitted 2016-08-04; First posted 2016-08-11 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-06

CONDITIONS: Hypotension
Keywords: Spinal anaesthesia
MeSH Terms: conditions — Hypotension | interventions — Anesthesia, Spinal; Ondansetron; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Ondansetron (Experimental)
  Interventions: Procedure: Spinal anaesthesia; Drug: Ondansetron
- Saline solution (Placebo Comparator)
  Interventions: Procedure: Spinal anaesthesia; Other: saline solution

INTERVENTIONS:
Procedure: Spinal anaesthesia
Drug: Ondansetron
  Arms: Ondansetron
Other: saline solution
  Arms: Saline solution

SUMMARY:
The intravenous injection of 8mg of ondansetron (a serotonin type 3 receptor antagonist) before spinal anaesthesia for caesarean section, leads to a smaller reduction in systolic arterial pressure (SAP).

The expected results are a decrease in the frequency and severity of hypotension, thus leading to improved comfort for the mother and decreased maternal and foetal morbidity. Indeed, episodes of hypotension are responsible for impaired foeto-placental circulation, with sometimes severe consequences for neonates.

It has been established that episodes of hypotension alter foetal pH. Investigators therefore hope to see a smaller reduction in SAP in the ondansetron group, and show a benefit for the infant.

One of the objectives of this study is also to observe a decrease in the quantity of vasopressors used and thus to avoid the adverse effects of their use in high doses.

The expected results are thus an improvement in haemodynamic stability during spinal anaesthesia for caesarean section.

The originality of this project lies in the use of a CNAP monitor (Continuous Non-invasive Arterial Pressure) as the collection of haemodynamic data will allow greater precision with the continuous measurement of AP, as well as a study of maternal cardiac output.

ELIGIBILITY:
Inclusion Criteria:

* Persons who have provided written informed consent
* Persons with national health insurance cover
* Patients aged over 18 years, ASA I or II
* About to undergo scheduled or non-scheduled caesarean section under spinal anaesthesia

Exclusion Criteria:

* Adults under guardianship
* Contra indication for spinal anaesthesia (SA) (refusal, haemodynamic instability, innate or acquired coagulation disorder)
* History of hypersensitivity to Zophren or local anaesthetics
* Heart and/or kidney failure
* Treatment with angiotensin converting enzyme (ACE) inhibitor, Beta Blockers, or angiotensin II receptor antagonist (ARA II), Zophren, atropine, Selective Serotonin Reuptake Inhibitors, Triptans
* Caesarean in a context of extreme emergency, with a time to foetal extraction incompatible with SA and the injection of Zophren, (up to 30 minutes) and requiring consent in an emergency.
* Pregnancy-related arterial hypertension (AHT)
* Pre-eclampsia
* Gestational diabetes

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-03; Primary Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
number of Systolic blood pressure below 90 mmHg | every 2 minutes from the intrathecal injection for 20 minutes, and then every 5 minutes until the end of the surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France